CLINICAL TRIAL: NCT04150302
Title: Development and Validation of a Questionnaire to Measure the Impact of Short Bowel Syndrome (SBS) and Its Treatments on Patients' Lives
Brief Title: Development and Validation of a Questionnaire to Measure the Impact of SBS and Its Treatments on Patients' Lives
Acronym: ARTEMIS_GC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Beaujon Hospital (Other); Société Francophone Nutrition Clinique et Métabolisme (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-A02034-53
Record Dates: First submitted 2019-09-23; First posted 2019-11-04 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-09

CONDITIONS: SBS - Short Bowel Syndrome
MeSH Terms: conditions — Short Bowel Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Exploratory interviews — Exploratory interviews to generate an interview guide
Other: Semi-directive interviews — Semi-directive interviews to collect qualitative data that will be used for questionnaire item generation
Other: Delphi Process — Cotation of newly developed items pertinence on a 4 points likert scale.
Other: Think aloud interviews — Debriefing session for the newly developed items: final possibility to adjust the tool before validating the psychometric proprieties of the questionnaire.
Other: Psychometric validation — Psychometric properties study

SUMMARY:
Today, patients express a very strong need to take into account the consequences of their disease and its treatments in their therapeutic follow-up. It is therefore essential to better understand the needs, expectations and values of patients with SBS in order to better understand the impact of the disease on their lives, and thus improve the conditions for medical, social, psychological and technical care. The clinical expertise of health professionals and meetings with patient associations demonstrate the major gap between the parameters taken into account by physician to evaluate the evolution of the SBS and the day-to-day experience of the disease perceived by the patient.

The objective of the ARTEMIS-GC study is to develop and validate an instrument to measure the impact of SBS and its treatments on daily life from the perspective of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with SBS defined by a hail length remaining in post-duodenal < 2 meters
* Patients with intestinal insufficiency, i.e. chronic malabsorption requiring energetic and/or hydro-electrolytic intravenous support for more than 6 months
* Patients with a period of at least 6 months after the establishment of the SBS
* Patients who has already had a return home after the establishment of the SBS for a period of at least 3 months

Exclusion Criteria:

* Patients with intestinal insufficiency but with a cause other than SBS
* Lack of understanding of the study
* Not speaking French

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years with SBS for more than 6 months and returned home for at least 3 months.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Scale calibration of the new developped questionnaire | about 30 minutes
  Calibration measure
Structure of the new developped questionnaire | about 30 minutes
  Structure identification
Convergence proprieties of the new developped questionnaire | about 30 minutes
  Convergence evaluation
Reproducibility of the new developped questionnaire | Up to 8 days
  Test of reproducibility

CONTACTS AND LOCATIONS:
Locations (1):
- Beaujon Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided